CLINICAL TRIAL: NCT05195463
Title: Comparison of the Efficiency of Abdominal Corset and Core Stabilization Exercises in the Treatment of Postpartum Diastasis Recti Abdominis
Brief Title: Efficiency of Abdominal Corset and Core Stabilization Exercises in the Treatment of Postpartum Diastasis Recti Abdominis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, merve yilmaz menek, Principle Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Merveylmz.
Record Dates: First submitted 2022-01-04; First posted 2022-01-19 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Diastasis Recti
Keywords: diastasis recti abdominis; core stabilization exercise; physiotherapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not know which group they belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First group (Experimental): Core stabilization exercises
  Interventions: Other: Exercise intervention
- Second group (Experimental): Combination of core stabilization and abdominal corset
  Interventions: Other: Exercise intervention by wearing abdominal corset
- Third group (Experimental): Only abdominal corset
  Interventions: Other: Corset intervention

INTERVENTIONS:
Other: Exercise intervention — Women with diastasis recti abdominis will do core stabilization exercises for the transversus abdominis muscle with 10 repetitions 3 days a week for 8 weeks. The exercises include diaphragmatic breathing exercises, core stabilization exercises for the transversus abdominis muscle, and pelvic floor contractions
  Arms: First group
Other: Exercise intervention by wearing abdominal corset — In this group, in addition to the first group, core stabilization exercises will be performed by wearing an abdominal corset. Participants will be asked to wear their corsets while performing their exercises.
  Arms: Second group
Other: Corset intervention — Participants included in this group will be required to wear only this corset all day (except for the bathroom) for 8 weeks.
  Arms: Third group

SUMMARY:
Participants will be randomly divided into three groups as core stabilization group, combination of core stabilization and corset group and only corset group.

DETAILED DESCRIPTION:
30 volunteer women who were diagnosed with diastasis recti abdominis by an obstetrician in Çamlıca Medipol Hospital, aged between 18-35 and met the inclusion criteria will be included in the study. Participants will be randomly divided into three groups. Participants in the first group will do core stabilization exercises for the transversus abdominis muscle 3 days a week for 8 weeks with 10 repetitions. In the second group, in addition to the first group, core stabilization exercises will be performed by wearing an abdominal corset. Participants included in the third group will be asked to wear only this corset all day (except for the bathroom) for 8 weeks. Anthropometric measurements, ultrasonographic evaluation, Visual Analogue Scale (VAS), Edinburgh Postnatal Depression Scale, abdominal muscle strength and endurance, Oswestry Disability Index will be evaluated as pretest and posttest.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 20-35,
* Having a normal birth,
* Being at least 6 weeks postpartum when DRA is diagnosed,
* Absence of any musculoskeletal or neurological problems,
* Volunteering to do the exercises

Exclusion Criteria:

* Cesarean delivery,
* Edinburgh Postnatal Depression questionnaire result being >13,
* Having a systemic disorder

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Enrollment: 45 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Ultrasanografic measurement | 5 minutes
  The distance between the rectus muscles will be measured by the obstetrician with ultrasound.
Visual Analogue Scale for pain assessment | 3 minutes
  The line has a value of 0 at the beginning and a value of 10 at the end. The patient is asked to indicate the intensity of the pain at rest or during activity. A value of 0 means no pain, a value of 10 means excruciating pain.
Abdominal muscle strength measurement | 5 minutes
  The abdominal muscle strength of the participants will be graded from 0 to 5 using manual muscle testing.
Abdominal muscle undurance measurement | 5 minutes
  n the measurement of muscle endurance, the participants will be asked to stand as long as they can in their position during the muscle strength measurement.
Edinburgh Postnatal Depression Scale | 5 minutes
  The scale is used to determine the risk of depression in the postpartum period and to measure the change in level and severity. Minimum value is 0 and maximum value is 30. Cut-off score of 13 is used to distinguish depressed from nondepressed women. High scores means worse outcomes.
Oswestry Disability Index for assesment of pain and quality of life | 5 minutes
  It is a questionnaire evaluating individuals' participation in activities of daily living due to low back pain.

SECONDARY OUTCOMES:
Weight measurement | 2 minutes
  Weight measurement in kilograms will be recorded with weighing machine.
Height measurement | 2 minutes
  Height measurement in meters will be recorded with tape measure

CONTACTS AND LOCATIONS:
Overall Officials: MERVE YILMAZ MENEK, Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will publish a manuscript about the result of this study for sharing results of the data with other researchers.